CLINICAL TRIAL: NCT00419003
Title: Continuation Riluzole in the Prevention of Relapse Following Ketamine in Major Depression
Brief Title: Research Study for Major Depressive Disorder: Investigation of Glutamate Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Sanjay Johan Mathew, MD, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-0850; 5M01RR000071-46 (NIH)
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lamotrigine; Ketamine; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine Pre-Treatment (Experimental): Patients who met enrolment criteria for phase 1 were randomly allocated to lamotrigine or placebo by a permuted block procedure consisting of blocks of two or four patients. The randomization list was created by a biostatistician with no patient contact. 300 mg of lamotrigine 2 hrs prior to ketamine infusion. Responders were randomized to one of two continuation pharmacotherapy groups, receiving either two capsules of riluzole 50 mg each (100 mg/d) or matching pill placebo under double-blind conditions.
  Interventions: Drug: Lamotrigine; Drug: Ketamine; Drug: Riluzole
- Placebo Pre-Treatment (Placebo Comparator): 2 hours prior to ketamine infusion each patient received three capsules of placebo identical in size, weight, appearance, and taste to the lamotrigine tablets. Responders were randomized to one of two continuation pharmacotherapy groups, receiving either two capsules of riluzole 50 mg each (100 mg/d) or matching pill placebo under double-blind conditions.
  Interventions: Drug: Ketamine; Drug: Riluzole

INTERVENTIONS:
Drug: Lamotrigine — anticonvulsant medication
  Other Names: lamictal
  Arms: Lamotrigine Pre-Treatment
Drug: Ketamine — subanesthetic dose of NMDAR antagonist
  Other Names: ketalar
Drug: Riluzole — glutamate release inhibitor
  Other Names: rilutek

SUMMARY:
This study is examining the safety and effectiveness of two medications, ketamine and riluzole, in treating patients with treatment resistant major depressive disorder. This study will also examine the effectiveness of an FDA approved drug called lamotrigine in decreasing the potential side effects associated with ketamine.

DETAILED DESCRIPTION:
This research proposal will investigate a glutamate-modulating agent, riluzole, in treatment-resistant patients who exhibit an acute, sustained response to a single dose of intravenous (IV) racemic ketamine. Fifty ketamine-responders will be randomized to riluzole or placebo in a 4-week, randomized, double-blind, continuation-phase study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21- 70 years of age
2. Subjects have a history of at least one previous episode of depression prior to the current episode (recurrent major depressive disorder) or have chronic major depressive disorder (at least two years' duration)
3. Subjects have not responded to an adequate trial of one antidepressant in the current episode

Exclusion Criteria:

1. Female subjects who are either pregnant or nursing
2. Serious, unstable illnesses
3. Any previous use or treatment with ketamine, or riluzole
4. Past intolerance to lamotrigine, including drug rash

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mathew, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Derived] Price RB, Nock MK, Charney DS, Mathew SJ. Effects of intravenous ketamine on explicit and implicit measures of suicidality in treatment-resistant depression. Biol Psychiatry. 2009 Sep 1;66(5):522-6. doi: 10.1016/j.biopsych.2009.04.029. Epub 2009 Jul 9. PMID 19545857
- [Derived] Mathew SJ, Murrough JW, aan het Rot M, Collins KA, Reich DL, Charney DS. Riluzole for relapse prevention following intravenous ketamine in treatment-resistant depression: a pilot randomized, placebo-controlled continuation trial. Int J Neuropsychopharmacol. 2010 Feb;13(1):71-82. doi: 10.1017/S1461145709000169. Epub 2009 Mar 17. PMID 19288975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intent-to-treat sample (n=26) was recruited from media/internet advertising (14), psychiatrist referral (8), or self-referral from the New York Mood Disorders Support Group (4). Patients had marked depressive severity, chronicity, and anxiety comorbidity, and were highly pharmacotherapy-resistant.
Pre-assignment Details: 2-wk psychotropic medication washout period (4 wk for fluoxetine)
Groups:
- Lamotrigine Pre-Treatment (Phase I)/Riluzole (Phase II); Placebo Pre-Treatment (Phase I)/Placebo (Phase II): Patients who met enrolment criteria for phase 1 were randomly allocated to lamotrigine or placebo by a permuted block procedure consisting of blocks of two or four patients. The randomization list was created by a biostatistician with no patient contact. Following baseline ratings, 2 h prior to i.v. ketamine infusion, patients received 300 mg lamotrigine or placebo by mouth. All non responders were exited from the study. All responders (in both the lamotrigine and placebo pre-treatment groups were treated as one group and randomized into either treatment with riluzole or placebo for Phase II)
Period: Phase I, Ketamine Infusion
Arm/Group | Lamotrigine Pre-Treatment (Phase I)/Riluzole (Phase II) | Placebo Pre-Treatment (Phase I)/Placebo (Phase II)
Started | 13 | 13
Completed | 7 | 7
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 6 | 6
Period: Phase 2, Riluzole/Placebo Follow-Up
Arm/Group | Lamotrigine Pre-Treatment (Phase I)/Riluzole (Phase II) | Placebo Pre-Treatment (Phase I)/Placebo (Phase II)
Started | 6 (14 completers of phase I didn't split up evenly (same way as phase I) in the riluzole/placebo phase.) | 8 (14 completers of phase I didn't split up evenly (same way as phase I) in the riluzole/placebo phase.)
Completed | 5 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine Pre-Treatment; Placebo Pre-Treatment: Patients who met enrolment criteria for phase 1 were randomly allocated to lamotrigine or placebo by a permuted block procedure consisting of blocks of two or four patients. The randomization list was created by a biostatistician with no patient contact. Following baseline ratings, 2 h prior to i.v. ketamine infusion, patients received 300 mg lamotrigine or placebo by mouth.
- Total: Total of all reporting groups
Arm/Group | Lamotrigine Pre-Treatment | Placebo Pre-Treatment | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.8) | 48.2 (11.8) | 48.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MARDS) Score (Acute Response to IV Ketamine in Patients With Treatment Resistant Major Depression)
Description: Montgomery-Asberg Depression Rating Scale, each of the ten items can be scored from 0 (absence of symptoms to 6 most severe) and has a total score range of 0-60. A lower score on a MADRS indicates a less severe depression. The primary outcome for the initial phase of the trial was the 24-h MADRS score, which included all 10 MADRS items.
Time Frame: 24 Hours
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Riluzole Group: Patients who responded (n=14) to the ketamine infusion (in either the lamotrigine or placebo pre-treatment groups) were randomized into phase II for treatment with either riluzole or placebo. One patient in the riluzole group was discontinued/withdrew consent before completing the study.
- Placebo: Patients who responded (n=14) to the ketamine infusion (in either the lamotrigine or placebo pre-treatment groups) were randomized into phase II for treatment with either riluzole or placebo.
Arm/Group | Riluzole Group | Placebo
Number analyzed (Participants) | 13 | 13
scores on a scale | 24.4 [15.9 to 33.0] | 22.0 [14.9 to 29.1]

2. Other Pre Specified Outcome: Efficacy of Lamotrigine in Decreasing IV Ketamine Psychotomimetic Side Effects
Description: Response rate and side effect differences to IV ketamine infusion based on lamotrigine and placebo pretreatment groups
Time Frame: 24, 48, or 72-hrs
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Riluzole Group; Placebo; Lamotrigine Pre-Treatment; Placebo Pre-Treatment: Patients who met enrolment criteria for phase 1 were randomly allocated to lamotrigine or placebo by a permuted block procedure consisting of blocks of two or four patients. The randomization list was created by a biostatistician with no patient contact. Following baseline ratings, 2 h prior to i.v. ketamine infusion, patients received 300 mg lamotrigine or placebo by mouth.
- Ketamine: IV infusion of 0.5 mg/kg of Ketamine Hydrochloride
Arm/Group | Riluzole Group | Placebo | Ketamine | Lamotrigine Pre-Treatment | Placebo Pre-Treatment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/26 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/6 | 5/8 | 26/26 | 5/13 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole Group (N=6) | Placebo (N=8) | Ketamine (N=26) | Lamotrigine Pre-Treatment (N=13) | Placebo Pre-Treatment (N=13)
Headache (Nervous system disorders) | 2 (6) | 0 (0) | 26 (26) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 3 (3) | 26 (26) | 0 | 0
Fatigue (Nervous system disorders) | 3 (3) | 2 (2) | 0 | 5 (5) | 0

LIMITATIONS AND CAVEATS:
The open-label administration of ketamine limits interpretation of phase 1 results. The sample size was too small to detect moderators and mediators of response. Third,lack of placebo-controlled efficacy data supporting riluzole's use in depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No